CLINICAL TRIAL: NCT03089905
Title: Neurodevelopmental Outcome After Standard Dose Sevoflurane Versus Low-dose Sevoflurane/Dexmedetomidine/Remifentanil Anaesthesia in Young Children- The TREX Trial
Brief Title: A Study to Compare the Long-term Outcomes After Two Different Anaesthetics
Acronym: TREX
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Sydney Children's Hospitals Network (Other); Baylor College of Medicine (Other); Boston Children's Hospital (Other); The Cleveland Clinic (Other); University of Texas, Southwestern Medical Center at Dallas (Other); Royal Children's Hospital (Other); Children's Hospital of Philadelphia (Other); Queensland Children's Hospital (Other Government); Perth Children's Hospital (Unknown); Women and Children's Hospital (Unknown); Istituto Giannina Gaslini (Other); Flinders Medical Centre (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TREX TRIAL; 2024-512385-34-00 (EU CTIS Number)
Record Dates: First submitted 2017-03-08; First posted 2017-03-24 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Anesthesia; Neurotoxicity; Child Development
MeSH Terms: conditions — Neurotoxicity Syndromes | interventions — Sevoflurane; Remifentanil; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Participants will be randomised to receive either low-dose sevoflurane/dexmedetomidine/remifentanil OR standard dose sevoflurane anaesthesia.
Who Masked: Outcomes Assessor
Masking Description: Randomisation 1:1 will be stratified by site and age at exposure (less than 12 months and greater than or equal to 12 months). Randomisation will be in blocks of variable size. The treating anaesthetist will not be blinded to treatment arm. The assessing neuropsychologist and parents will be blinded to treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sevoflurane/dexmedetomidine/remifentanil (Experimental): Dexmedetomidine: loading dose of 1mcg/kg over 10 minutes followed by an infusion of at 1 mcg/kg/hr.
  Remifentanil: loading dose 1 mcg/kg over 2 minutes followed by an infusion starting at 0.1 mcg/kg/min or greater.
  Sevoflurane: end tidal concentration of 0.6 -0.8% or less.
  Interventions: Drug: Sevoflurane; Drug: Remifentanil; Drug: Dexmedetomidine
- Sevoflurane (Active Comparator): End tidal concentration of 2.5-3.0% or greater.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane — Experimental arm: end tidal concentration of 0.6 -0.8% or less. Active comparator arm: end tidal concentration of 2.5-3.0% or greater.
  Other Names: Sevorane
Drug: Remifentanil — Experimental arm: loading dose: 1 mcg/kg, infusion starting at 0.1 mcg/kg/min or greater.
  Other Names: Ultiva
  Arms: Sevoflurane/dexmedetomidine/remifentanil
Drug: Dexmedetomidine — Experimental arm: loading dose:1mcg/kg, infusion: 1 mcg/kg/hr.
  Other Names: Precedex; Dexmedetomidine Ever Pharma
  Arms: Sevoflurane/dexmedetomidine/remifentanil

SUMMARY:
There is considerable evidence that most general anaesthetics modulate brain development in animal studies. The impact is greater with longer durations of exposure and in younger animals. There is great controversy over whether or not these animal data are relevant to human clinical scenarios.

The changes seen in preclinical studies are greatest with GABA agonists and NMDA antagonists such as volatile anaesthetics (eg sevoflurane), propofol, midazolam, ketamine, and nitrous oxide. There is less evidence for an effect with opioid (such as remifentanil) or with alpha 2 agonists (such as dexmedetomidine).

Some, but not all, human cohort studies show an association between exposure to anaesthesia in infancy or early childhood and later changes in cognitive tests, school performance or risk of developing neurodevelopmental disorders. The evidence is weak due to possible confounding.

A recent well designed cohort study (the PANDA study) comparing young children that had hernia repair to their siblings found no evidence for a difference in a range of detailed neuropsychological tests. In that study most children were exposed to up to two hours of anaesthesia. The only trial (the GAS trial) has compared children having hernia repair under regional or general anesthesia and has found no evidence for a difference in neurodevelopment when tested at two years of age. The GAS and PANDA studies confirm the animal data that short exposure is unlikely to cause any neurodevelopmental impact.

The impact of longer exposures is still unknown. In humans the strongest evidence for an association between surgery and poor neurodevelopmental outcome is in infants having major surgery. However, this is also the group where confounding is most likely.

The aim of our study is to see if a new combination of anaesthetic drugs results in a better long-term developmental outcome than the current standard of care for children having anaesthesia expected to last 2 hours or longer.

Children will be randomised to receive either a low dose sevoflurane/remifentanil/dexmedetomidine or standard dose sevoflurane anaesthetic.

They will receive a neurodevelopmental assessment at 3 years of age to assess global cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Younger than 2 years (chronological age)
* Scheduled for anaesthesia that is expected to last at least 2 hours (and/or total operating room time is scheduled to be at least 2.5 hours)
* Has a legally acceptable representative capable of understanding the informed consent document and providing consent on the participant's behalf.

Exclusion Criteria:

* Known neurologic, chromosomal or congenital anomaly which is likely to be associated with poor neurobehavioural outcome
* Existing diagnosis of behavioural or neurodevelopmental disability
* Prematurity (defined as < 36 weeks gestational age at birth)
* Birth weight less than 2 kg.
* Congenital cardiac disease requiring surgery
* Intracranial neurosurgery and intracranial craniofacial surgery (isolated cleft lip is not an exclusion)
* Previous cumulative exposure to general anaesthesia exceeding 2 hours
* Planned future cumulative exposure to anaesthesia exceeding 2 hours before the age of 3 years.
* Any specific contra-indication to any aspect of the protocol
* Previous adverse reaction to any anaesthetic
* Circumstances likely to make long term follow-up impossible
* Living in a household where the primary language spoken at home is not a language in which we can administer the Wechsler Preschool and Primary School Intelligence Scale
* Planned postoperative sedation with any agent except opioids (e.g. benzodiazepines, dexmedetomidine, ketamine, barbiturates, propofol, clonidine, chloral hydrate, and other non-opioid sedatives). For example if such sedation is planned for post-operative ventilation

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 450 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Full Scale IQ | 3 years of age
  Global cognitive function as assessed by the full scale IQ score of the Wechsler Preschool and Primary School Intelligence Scale.

SECONDARY OUTCOMES:
incidence of intra-operative hypotension | 150 minutes- duration of surgery (baseline)
  Blood pressure measurements will be recorded during surgery
incidence of intra-operative bradycardia | 150 minutes- duration of surgery (baseline)
  Heart rate will be recorded during surgery
Post-operative pain | 60 minutes- after surgery
  Pain scores will be recorded after surgery
Time to recovery | 60 minutes- after surgery
  Time of removal of airway, eye-opening and discharge from PACU will be recorded.
Language outcomes | 3 years of age
  Clinical Evaluation of Language Fundamentals- Preschool, Version 2 (CELF-P2)
Attention/Executive Function/impulse control | 3 years of age
  A Developmental NEuroPSYchological Assessment- Second Edition (NEPSY-2): Statue Subtest
Memory | 3 years of age
  A Developmental NEuroPSYchological Assessment- Second Edition (NEPSY-2): Narrative memory
Adaptive behaviour | 3 years of age
  Adaptive Behavior Assessment System - Third Edition (ABAS-III)
Clinical Behavior | 3 years of age
  Child Behavior Checklist (CBCL)
Executive Function | 3 years of age
  Behavior Rating of Executive Function- Preschool (BRIEF-P)
Social Skills | 3 years of age
  Social Skills Improvement System (SSIS)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Davidson, MD, Study Chair — Royal Children's Hospital
Locations (21):
- United States (5):
  - Boston Children's Hospital, Boston, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
- Australia (7):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, Brisbane, Queensland
  - Women's and Children's Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Royal Children's Hospital, Parkville, Victoria
  - Perth Children's Hospital, Perth, Western Australia
- Italy (8):
  - Presidio Ospedale Infantile C.Arrigo Azienda Ospedaliera, Alessandria
  - Azienda ospedaliero-universitaria di Bologna, Bologna
  - Azienda Ospedaliero-Universitaria Meyer, Florence
  - Istituto Giannina Gaslini, Genova
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico - Clinica Mangiagalli, Milan
  - Vittore Buzzi Children's Hospital, Milan
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Ospedale Bambino Gesù, Roma
- La Paz University Hospital, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data set collected for this analysis of the TREX trial will be available six months after publication of the primary outcome.
  The study protocol, analysis plan and consent forms will also be available. The data may be obtained from the Murdoch Children's Research Institute by emailing andrew.davidson@rch.org.au.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publication of primary outcome
Access Criteria: Prior to releasing any data the following are required: a data access agreement must be signed between relevant parties, the TREX Trial Steering Committee must see and approve the analysis plan describing how the data will be analysed, there must be an agreement around appropriate acknowledgement and any additional costs involved must be covered. Data will only be shared with a recognised research institution which has approved the proposed analysis plan.

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/05/NCT03089905/SAP_000.pdf